CLINICAL TRIAL: NCT06558656
Title: A Randomized, Open Label, Two Sequence, Two Period, Double Crossover-design Phase I Clinical Trial of NTQ5082 Capsules Taken by Healthy Subjects on an Empty Stomach (i.e, Fasting) as Well as After a Meal (i.e. Fed)
Brief Title: Effect of Food of NTQ5082 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NTQ5082-24102
Record Dates: First submitted 2024-07-23; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Complement-mediated Hemolytic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting-Fed (Experimental): Fasting-Fed
  Interventions: Drug: NTQ5082 capsule
- Fed-Fasting (Experimental): Fed-Fasting
  Interventions: Drug: NTQ5082 capsule

INTERVENTIONS:
Drug: NTQ5082 capsule — Part 1:The subjects are orally administered NT5082 capsules on an empty stomach in the first cycle and after a meal in the second cycle.
  Part 2:The subjects are orally administered NT5082 capsules after a meal in the first cycle and on an empty stomach in the second cycle.

SUMMARY:
NTQ5082 capsule is a small molecule CFB factor inhibitor. The study is a randomized, open label, two sequence, two period, double crossover-design phase 1 clinical trial to evaluate the food effect on PK after a single oral administration of NTQ5082 capsules and the safety and tolerability of single oral administration of NTQ5082 capsules on an empty stomach (i.e, fasting) as well as after a meal (i.e. fed) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, ≥18 years and ≤45 years in age.
2. 19.0 kg/m2≤BMI≤26.0 kg/m2, and male weight must be ≥50 kg, female weight must be ≥45 kg;
3. Those who sign an informed consent form before the experiment and fully understand the content, process, and possible adverse reactions of the experiment;
4. The subjects are able to communicate well with the researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Participants who have participated in any other drug clinical trials and used the investigational drug within 3 months prior to the trial;
2. Individuals who have chronic or active gastrointestinal diseases such as esophageal disease, gastritis, gastric ulcer, gastroesophageal reflux, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery within the past three years, and who are still clinically significant according to researchers;
3. Individuals with clear diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, metabolic disorders, etc. that require medical intervention or other diseases that are not suitable for clinical trials (such as a history of mental illness);
4. Known or suspected history of immunodeficiency (such as frequent recurrent infections), genetic or acquired complement deficiency;
5. There is a clear history of capsule microbial infection within the first 6 months of screening; Including but not limited to: history of infection with Streptococcus pneumoniae, Bacillus anthracis, Salmonella, Salmonella typhi, Klebsiella pneumoniae, Pseudomonas aeruginosa, Bacteroides fragilis, Neisseria meningitidis, Haemophilus influenzae, Legionella pneumophila;
6. Individuals with a history of tuberculosis infection or currently suffering from tuberculosis infection;
7. Active systemic bacterial, viral, or fungal infection within 14 days prior to administration;
8. Fever (≥ 38 ℃) occurred within 7 days before administration;
9. Individuals with a history of allergies to experimental preparations, any of their components or related preparations, or to drugs, food or other substances;
10. Those who cannot tolerate venous puncture or have a history of dizziness or needle fainting;
11. Patients who have undergone surgery within 6 months prior to the use of the investigational drug, as determined by the researcher, that may affect drug absorption, distribution, metabolism, and excretion; Or have undergone surgical procedures within 4 weeks prior to using the investigational drug; Or those who plan to undergo surgical procedures during the trial period;
12. Those who have used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, traditional Chinese patent medicines and simple preparations and dietary supplements) within 2 weeks before using the study drug; Or screen for drugs with a duration of less than 5 half lives (whichever is longer);
13. Individuals who have received the vaccine or live attenuated vaccine within 14 days prior to using the investigational drug, or who plan to receive the vaccine during the trial period;
14. Individuals with QTc>450 milliseconds (male) or QTc>470 milliseconds (female) during screening;
15. Individuals who have donated blood or experienced significant blood loss (>400mL) within 3 months prior to the use of the investigational drug, those who have received blood transfusions or used blood products, or those who intend to donate blood or blood components during or within 3 months after the end of the trial;
16. Drug abusers or those who have used soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine, etc.) within the past year before using research drugs; Or those who test positive for urinary toxicity screening;
17. Smokers or those who have smoked more than 5 cigarettes per day in the 3 months prior to using the study drug, or those who cannot stop using any tobacco products during the trial period;
18. Alcoholics or frequent drinkers within the 6 months prior to the experiment, who consume more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Those who are unwilling to stop drinking alcohol or any alcoholic products during the trial period; Or those who test positive for alcohol breath test;
19. Individuals who consume excessive amounts of tea, coffee, and/or caffeinated beverages (8 or more cups, 1 cup=250 mL) daily, or who do not agree to stop drinking tea, coffee, and/or caffeinated beverages during the trial period;
20. Individuals who consume a diet (including grapefruit or grapefruit products, etc.) that may affect the metabolism of the investigational drug within 7 days prior to use, or who are deemed by the researcher to have other diets that may affect the absorption, distribution, metabolism, or excretion of the drug, or who do not agree to stop consuming the aforementioned foods during the trial period;
21. Those who have special dietary requirements and cannot follow a uniform diet;
22. Female subjects are pregnant or breastfeeding women; Or engaging in unprotected sexual activity within 2 weeks prior to the use of the investigational drug; Those who have used oral contraceptives within 30 days prior to the use of the study drug, or those who have used long-acting estrogen or progesterone injections or implants within 6 months prior to the use of the study drug;
23. If the subject (or their partner) has a pregnancy plan, sperm and egg donation plan, or is unwilling to take one or more non pharmacological contraceptive measures (such as complete abstinence, contraceptive rings, partner ligation, etc.) within 3 months after the last dose of medication from the time of signing the informed consent form;
24. Physical examination, electrocardiogram, abdominal ultrasound, chest radiograph, laboratory tests (blood routine, reticulocyte count, procalcitonin, high-sensitivity C-reactive protein, urine routine, blood biochemistry, thyroid function, coagulation function, D-dimer, blood transfusion, blood pregnancy), vital signs, and clinically significant abnormalities in various examinations (subject to the judgment of the research doctor);
25. Participants may not be able to complete this study due to other reasons or may have other reasons deemed inappropriate by the researchers to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
AUC0-last | up to 15 days
AUC0-∞ | up to 15 days
Cmax | up to 15 days
Tmax | up to 15 days
t1/2 | up to 15 days
CL/F | up to 15 days
Vz/F | up to 15 days

SECONDARY OUTCOMES:
the safety and tolerability | up to 15 days
  Safety and tolerability as assessed through collection of Adverse Event, Serious Adverse Event, Clinical Chemistry/Haematology/Coagulation/Vital Signs and ECG

CONTACTS AND LOCATIONS:
Locations (1):
- The Third hospital of Changsha, Changsha, Hunan, China